CLINICAL TRIAL: NCT00990951
Title: Double-blind, Randomized, Placebo-controlled Study of Efficacy of Association of Senna Alexandrina, Cassia Fistula, Tamarindus Indica, Coriandrum Sativum, Periandra Mediterranea in Patients With Functional Intestinal Constipation
Brief Title: Study of Efficacy of Association of Senna Alexandrina Mill and Associations on Functional Intestinal Constipation
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was interrupted by recruitment failure.
Sponsor: Marjan Industria e Comercio ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJ 3001-09
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Sennosides; Association

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Senna alexandrina and associations (Experimental): Association of Senna alexandrina Mill (sena), Cassia fistula L., Tamarindus indica L., Coriandrum sativum L., Periandra mediterranea Taub
  Interventions: Drug: Senna alexandrina and associations

INTERVENTIONS:
Drug: Senna alexandrina and associations — Drugs: Senna alexandrina Mill (sena), Cassia fistula L., Tamarindus indica L., Coriandrum sativum L., Periandra mediterranea Taub
  1 tablet PO twice a day
  Other Names: Brand name: Tamaril

SUMMARY:
The purpose of this study is to evaluate the efficacy of association of Senna alexandrina Mill (sena), Cassia fistula L., Tamarindus indica L., Coriandrum sativum L., Periandra mediterranea Taub. in patients with functional constipation.

DETAILED DESCRIPTION:
This is a phase III trial, placebo-controlled with a parallel-group design.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-65 years with functional constipation by ROME IIII criteria
* In the opinion of the investigator the patient will adhere to the protocol
* Voluntary able to understand the nature and purpose of the study, including the risks and adverse effects and with intent to cooperate with the researcher and act in accordance with the requirements of the entire protocol, which was confirmed by signing the Consent Informed

Exclusion Criteria:

* hypersensitivity to any component
* pregnant or lactating
* abdominal pain of unknown etiology
* suspected intestinal occlusion and sub-occlusion
* suspected abdominal inflammatory conditions (as appendicitis, peritonitis, cystitis, endometritis)
* Crohn disease and colitis
* Suspected intestinal constipation due abdominal surgery, neurological disorders (as aganglionoses, Parkinson disease, medullar tumor, stroke, multiple sclerosis), systemic sclerosis, multiple myeloma, scleroderma
* Subjects with congenital mega colon, anorectal congenital malformation, inflammatory bowel disease or intestinal carcinoma
* history of mal-absorption diseases
* history of anemia, weight loss or anal bleeding
* history of hypothyroidism, hyperthyroidism and insulin-dependent diabetes mellitus
* known of positive result for human immunodeficiency virus test
* heart, liver, lung or kidney important condition
* drug or alcohol dependence
* knowledge or suspicion of malignancy
* body mass index < 18
* body mass index > 30
* participation on any experimental study 12 months prior this study
* familiar history of colon carcinoma or inflammatory disease
* Lack of adherence to the procedures of the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
average frequency of bowel movements measured at baseline and at 2 weeks of treatment | 2 weeks

SECONDARY OUTCOMES:
number of consecutive days that patients do not evacuate | 2 weeks
Proportion of stools with pain and difficulty | 2 weeks
degree of improvement of constipation according to the subjective evaluation of the volunteer, measured by the scores of the Global Assessment of the patient | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria EA Moraes, MD, PhD, Principal Investigator — Federal University of Ceara - UNIFAC
Locations (1):
- Departamento de Fisiologia e Farmacologia, Ceará, Fortaleza, Brazil